CLINICAL TRIAL: NCT03129178
Title: Beet the Cold: The Effect of Inorganic Nitrate Supplementation on Peripheral Blood Flow and Pain in Individuals With Raynaud's Phenomenon. A Pilot, Double-blind, Placebo Controlled, Randomised Crossover Trial
Brief Title: Beet the Cold: The Effect of Inorganic Nitrate Supplementation in Individuals With Raynaud's Phenomenon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Portsmouth (Other)
Collaborators: Loughborough University (Other); University of Exeter (Other)
Responsible Party: Principal Investigator, Ant Shepherd, Lecturer, University of Portsmouth
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2017-03-30; First posted 2017-04-26 (Actual); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2019-09

CONDITIONS: Raynaud Phenomenon
Keywords: Nitrate; Nitric oxide; Microvascular
MeSH Terms: conditions — Raynaud Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind, randomised control trial. Supplements will be dispensed by nurses or a member of the research team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beetroot juice then nitrate depleted beetroot juice (Experimental): Participants will be asked to consume 140ml of beetroot juice prior to their first experimental visit. Participants will then be asked to consume 70ml a day for 2 weeks and final visit the investigators once more following another 140ml drink.
  Interventions: Dietary Supplement: Concentrated beetroot juice
- Nitrate depleted beetroot juice then beetroot juice (Experimental): Participants will be asked to consume 140ml of placebo prior to their first experimental visit. Participants will then be asked to consume 70ml a day for 2 weeks and final visit the investigators once more following another 140ml drink.
  Interventions: Dietary Supplement: Concentrated beetroot juice

INTERVENTIONS:
Dietary Supplement: Concentrated beetroot juice — Acute and chronic supplementation of beetroot juice.

SUMMARY:
Individuals with Raynaud's phenomenon often experience episodes of reduced blood flow to their fingers and toes during times of stress or cold exposure, causing significant discomfort and pain. Typically, treatment for these individuals involves using drugs like Glyceryl Trinitrate (GTN), which increases blood flow to the fingers and toes by increasing a substance called nitric oxide in the blood. Unfortunately, repeated use of these drugs increases tolerance to them, meaning higher doses are required to produce the same effect. However, increasing the dose can cause more side effects like headaches, and is therefore not considered an ideal long-term therapy.

Leafy green vegetables, especially beetroot, contain high amounts of nitrate and are beneficial to blood vessel health, since nitrate from the diet can also be turned into the important blood vessel relaxer, nitric oxide. Unlike GTN, people don't appear to develop a tolerance to dietary nitrate or experience negative side effects.

Therefore, this study aims to see if short and longer term beetroot juice supplementation can improve blood flow to the hands and feet in individuals with Raynaud's phenomenon, as well as reduce their pain. This study will tell us how many people are needed for a definitive trial investigating whether beetroot juice can help treat Raynaud's phenomenon.

Raynaud's phenomenon can cause significant discomfort and pain to individuals. Dietary nitrate appears to offer a simple, low cost means of improving blood flow to the hands and feet which should reduce both the discomfort and pain experienced characterising this condition. This study will advance our understanding of the causes of Raynaud's phenomenon, specifically the role that the nitrate-nitrite-nitric oxide pathway might play in changing Raynaud's phenomenon symptoms and identifying targets for intervention.

DETAILED DESCRIPTION:
Raynaud's phenomenon (RP) is characterised by a recurrent transient vasospasm of the fingers or toes in response to a cold or stressful stimulus. Nitric oxide (NO•) is a known vasodilator and NO• donors, such as Glyceryl Trinitrate (GTN), improve blood flow in patients with RP and in cold sensitive individuals (Figure 1, see accompanying document). However, individuals develop a tolerance to GTN and show diminishing vasodilatory effects with chronic treatment. In addition, the deleterious side effects such as headaches means that organic nitrates (i.e. GTN and isosorbide mononitrate) are not optimal longterm therapies for RP. Alternative treatments therefore, warrant further investigation.

Diets rich in fruit and vegetables has been shown to be effective in reducing blood pressure. In addition, it lowers the risk of morbidity and mortality from cardiovascular disease and are thought to be beneficial to cardiovascular health due to their vasodilatory effects. As diet exhibits such tremendous intra- and inter-individual variation, elucidating which components of such a diet are responsible for this effect is difficult. There is a growing weight of evidence from both human and animal studies that nitrate and nitrite derived from the diet can serve as a source for nitric oxide (NO; please see below), particularly where it is deficient. Indeed, the greatest protective effect on cardiovascular disease is to be found in those diets with the greatest consumption of green leafy and or cruciferous vegetables which typically have high nitrate content.

NO is produced in the body in two ways. The first requires the availability the amino acid L-arginine, molecular oxygen, and families of enzymes, the nitric oxide synthases (NOS); that is the NOS pathway. The second pathway is independent of NOS pathway and involves the stepwise enzymatic and chemical reduction of inorganic nitrate to nitrite. A major source of nitrite in humans is the reduction of dietary nitrate by facultative anaerobic bacteria in the mouth. The remaining nitrite is then absorbed into the circulation where it acts as a storage pool for subsequent NO• production, which is expedited in hypoxaemia.

Localised hypoxemia such as that observed in the digital vasculature of individuals with RP is a potential therapeutic target for dietary nitrate supplementation. In contrast to organic nitrates (GTN), inorganic nitrate (in the form of beetroot juice) does not cause the same negative side effects or demonstrate tachyphylaxis whilst it does notable improve skin blood flow, microvascular function and lower blood pressure (BP) in healthy individuals and chronic conditions such as hypertension, peripheral arterial disease, heart failure and chronic obstructive pulmonary disease. Thus concentrated beetroot juice (CBJ) may offer an inexpensive, safe and potentially effective intervention to improve the pain and reduced peripheral blood flow characterising individuals with RP.

RP can cause significant discomfort and pain to individuals during a vasospasm. Dietary nitrate appears to offer a simple, low cost means of modifying blood flow to the peripheries and, ultimately, reducing both the discomfort and pain experienced by individuals with RP. This study will also advance our understanding of the aetiology and pathophysiology of RP, specifically the role that the nitrate-nitrite-nitric oxide pathway might play in modulating RP symptoms. An understanding of the effects of concentrated beetroot juice on microvascular blood flow and pain may lead to a range of simple, low cost and effective therapeutic interventions to prevent and treat episodes of RP.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged 18 years or above.
* Diagnosed with Raynaud's Phenomenon.
* Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* Patients with significant renal impairment (eGFR<30)
* Uncontrolled hypertension,
* Taking regular organic nitrates, nicorandil, or thiazolidinidiones,
* or any medication which may interfere with data interpretation or safety,
* who have had a myocardial infarction or cerebro-vascular event,
* who smoke,
* or any other serious medical condition which would interfere with data interpretation or safety will be excluded from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sport and Exercise Science, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to release IPD, until all avenues of further funding have been exhausted.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 96 people were assessed for eligibility from clinic letters, word of mouth, local groups and via the clinical trials website. Recruitment occurred from 06-07-2017 - 29-05-2018.
Pre-assignment Details: 27 participants were consented.
Groups:
- Beetroot Juice, Then Nitrate Depleted Beetroot Juice: Participants consumed 140ml of beetroot juice prior to their first experimental visit. Participants will then be asked to consume 70ml a day for 2 weeks and final visit the investigators once more following another 140ml drink.
  Following a 7 day washout, then swapped into the nitrate depleted beetroot juice arm.
- Nitrate Depleted Beetroot Juice, Then Beetroot Juice: Participants consumed 140ml of nitrate depleted beetroot juice prior to their first experimental visit. Participants will then be asked to consume 70ml a day for 2 weeks and final visit the investigators once more following another 140ml drink.
  Following a 7 day washout, then swapped into the beetroot juice arm.
Period: Overall Study
Arm/Group | Beetroot Juice, Then Nitrate Depleted Beetroot Juice | Nitrate Depleted Beetroot Juice, Then Beetroot Juice
Started | 13 | 13
Completed | 12 | 11
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Beetroot Juice, Then, Nitrate Depleted Beetroot Juice: Participants consumed 140ml of beetroot juice prior to their first experimental visit. Participants will then be asked to consume 70ml a day for 2 weeks and final visit the investigators once more following another 140ml drink.
  Following a 7 day washout, then swapped into the nitrate depleted beetroot juice arm.
- Nitrate Depleted Beetroot Juice, Then, Beetroot Juice: Participants consumed 140ml of nitrate depleted beetroot juice prior to their first experimental visit. Participants will then be asked to consume 70ml a day for 2 weeks and final visit the investigators once more following another 140ml drink.
  Following a 7 day washout, then swapped into the beetroot juice arm.
- Total: Total of all reporting groups
Arm/Group | Beetroot Juice, Then, Nitrate Depleted Beetroot Juice | Nitrate Depleted Beetroot Juice, Then, Beetroot Juice | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 7 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (16.0) | 63.0 (15.2) | 64.3 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 10 | 12 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Peripheral Blood Flow
Description: Peripheral blood flow (CVC = skin flux/MAP; flux.mmHg-1).
Time Frame: Baseline (day 1), Acute (2 or 23), Chronic (day 16 or 36).
Population: 20 individuals with raynauds phenomenon. Result reported is Blood flow (CVC), 10 minutes after rewarming for the chronic exposures (Baseline (day 1), visit 2 (day 2), 3 (day 16), 4 (day 23) and 5 (day 36) respectfully).
Measure: Mean (Standard Deviation); unit: flux.mmHg-1
Groups:
- Concentrated Beetroot Juice: Participants will be asked to consume 140ml of beetroot juice prior to their first experimental visit. Participants will then be asked to consume 70ml a day for 2 weeks and final visit the investigators once more following another 140ml drink.
  Concentrated beetroot juice: Acute and chronic supplementation of beetroot juice.
- Nitrate Depleted Beetroot Juice: Participants will be asked to consume 140ml of placebo prior to their first experimental visit. Participants will then be asked to consume 70ml a day for 2 weeks and final visit the investigators once more following another 140ml drink.
  Concentrated beetroot juice: Acute and chronic supplementation of beetroot juice.
Arm/Group | Concentrated Beetroot Juice | Nitrate Depleted Beetroot Juice
Number analyzed (Participants) | 20 | 20
flux.mmHg-1
  Baseline (day 1) | 3.7 (0.4) | 3.7 (0.4)
  Acute (2 or 23) | 4.1 (0.3) | 3.7 (0.3)
  Chronic (day 16 or 36) | 4.7 (0.4) | 5.2 (0.4)

2. Primary Outcome: Skin Temperature.
Description: Skin temperature (via thermal imaging).
Time Frame: Baseline (day 1), Acute (2 or 23), Chronic (day 16 or 36).
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Concentrated Beetroot Juice | Nitrate Depleted Beetroot Juice
Number analyzed (Participants) | 23 | 23
Degree Celsius
  Baseline (day 1) | 32.4 (3.0) | 32.4 (3.0)
  Acute (day 2 or 23) | 32.1 (2.9) | 32.0 (3.0)
  Chronic (day 16 or 36) | 32.2 (3.4) | 32.4 (2.9)

3. Secondary Outcome: Perceived Discomfort
Description: Perceived discomfort.
  Thermal discomfort were measured using a 20 cm scale (0 = very cold/uncomfortable; 10 = neutral; 20 = very hot/comfortable; modified from Zhang et al. (2004)) and recorded prior to immersion, during immersion and every 2 minutes of the rewarming period.
Time Frame: Baseline (day 1), Acute (2 or 23), Chronic (day 16 or 36).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Concentrated Beetroot Juice | Nitrate Depleted Beetroot Juice
Number analyzed (Participants) | 23 | 23
score on a scale
  Baseline (day 1) | 13.4 (3.8) | 13.4 (3.8)
  Acute (day 2 or 23) | 13.1 (3.2) | 12.6 (3.7)
  Chronic (day 16 or 36) | 13.5 (3.5) | 12.9 (3.0)

4. Secondary Outcome: Acceptability to Participants
Description: Interview. Specifically, semi-structured interviews explored participants' experiences of the study procedures and consumption of beetroot juice. Interviews were conducted by a researcher with experience in qualitative research methods. Interviews were recorded, transcribed verbatim, and analysed through thematic analysis as outlined by Braun and Clarke (2006). Participants were asked about the testing procedures and their thoughts on the juice.
Time Frame: During qualitative interviews after the intervention has ended (post day 36).
Measure: Count of Participants; unit: Participants
Arm/Group | Concentrated Beetroot Juice | Nitrate Depleted Beetroot Juice
Number analyzed (Participants) | 10 | 10
Participants | 10 | 10

5. Secondary Outcome: Overall Number of Participants Recruited
Description: Number of participants who remained in the study
Time Frame: From start of study recruitment until the last participant is randomised. Estimated assesment period 6 - 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Concentrated Beetroot Juice
Number analyzed (Participants) | 27
Participants | 23

6. Secondary Outcome: Perceived Pain
Description: Perceived pain.
  Pain sensation was assessed using a numerical rating scale for pain (0 no pain, 10 unimaginable, unspeakable pain; (Ferreira-Valente et al., 2011)) at the same time points.
Time Frame: Baseline (day 1), Acute (2 or 23), Chronic (day 16 or 36).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Concentrated Beetroot Juice | Nitrate Depleted Beetroot Juice
Number analyzed (Participants) | 23 | 23
score on a scale
  Baseline (day 1) | 0.2 (0.6) | 0.2 (0.6)
  Acute (day 2 or 23) | 0.3 (0.8) | 0.2 (0.6)
  Chronic (day 16 or 36) | 0.2 (0.6) | 0.9 (2.7)

7. Secondary Outcome: Feasible to Participants
Description: Feasible to participants via interview. Specifically, semi-structured interviews explored participants' experiences of the study procedures and consumption of beetroot juice. Interviews were conducted by a researcher with experience in qualitative research methods. Interviews were recorded, transcribed verbatim, and analysed through thematic analysis as outlined by Braun and Clarke (2006).
Time Frame: During qualitative interviews after the intervention has ended (post day 36).
Population: Qualitative outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Concentrated Beetroot Juice | Nitrate Depleted Beetroot Juice
Number analyzed (Participants) | 10 | 10
Participants | 10 | 10

8. Secondary Outcome: Establish Retention Rates
Description: Establish retention rates (Descriptive statistics)
Time Frame: From date of randomization until the end of the last study visit. Estimated assesment period 6 - 52 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Overall Number of Participants Analyzed: This Overall Number of Participants Analyzed reflects the total number of individuals approached for recruitment for this study
Arm/Group | Overall Number of Participants Analyzed
Number analyzed (Participants) | 27
Participants | 23

ADVERSE EVENTS:
Time Frame: Two weeks for each intervention.
Groups:
- Concentrated Beetroot Juice: Participants will be asked to consume 140ml of beetroot juice prior to their first experimental visit. Participants will then be asked to consume 70ml a day for 2 weeks and final visit the investigators once more following another 140ml drink.
  Concentrated beetroot juice: Acute and chronic supplementation of beetroot juice.
  Total time on this arm is 14 days.
- Nitrate Depleted Beetroot Juice: Participants will be asked to consume 140ml of placebo prior to their first experimental visit. Participants will then be asked to consume 70ml a day for 2 weeks and final visit the investigators once more following another 140ml drink.
  Concentrated beetroot juice: Acute and chronic supplementation of beetroot juice.
  Total time on this arm is 14 days.
Arm/Group | Concentrated Beetroot Juice | Nitrate Depleted Beetroot Juice
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 3/26 | 2/26
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concentrated Beetroot Juice (N=26) | Nitrate Depleted Beetroot Juice (N=26)
GI distress (Gastrointestinal disorders) | 1 (1) | 1 (1) — Reports of upset stomach
Nausea / sickness (General disorders) | 1 (1) | 1 (1) — Reports of sickness and nausea
Hot flush (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Reports of transient periods of hot flushes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/78/NCT03129178/Prot_SAP_000.pdf